CLINICAL TRIAL: NCT04630847
Title: An Open-Label Phase I Clinical Trial of Vancomycin Followed by Familial Fecal Microbiota Transplant in Adult Subjects With Autism Spectrum Disorder (ASD)
Brief Title: Familial Fecal Microbiota Transplant for the Treatment of Subjects With Autism Spectrum Disorders
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ProgenaBiome (Other)
Collaborators: Ventura Clinical Trials (Unknown); Microbiome Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCT-1
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: microbiome; dysbiosis; FMT; fecal transpant; fecal microbiota transplant
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Dysbiosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autism Subjects (Experimental): These subjects will be administered fecal microbiota transplant by colonoscopy
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — FMT utilizing stool from first degree relatives

SUMMARY:
This is an open-label clinical trial to evaluate the benefits of familial fecal microbiota transplant following a 6-week treatment with Vancomycin in adult subjects with ASD for treatment of social deficits and language delays.

DETAILED DESCRIPTION:
This is an open-label clinical trial to evaluate the benefits of familial fecal microbiota transplant following a 6-week treatment with Vancomycin in adult subjects with ASD for treatment of social deficits and language delays. Participants are given FMT by colonoscopy

ELIGIBILITY:
Inclusion Criteria:

1. Subject at least six years of age.
2. Subject has confirmed diagnosis of ASD based on the DSM-V.
3. Subject with ASD whose parents/caregiver/guardian/LAR can complete informed consent process.
4. A reliable parent or caregiver who can report the side effects and communicate effectively with the research team.
5. Comorbid gastrointestinal symptoms
6. Stable medications during the two months prior to enrollment.
7. Currently receiving interventions in the community or school for ASD.
8. If female and of childbearing potential, must be willing to utilize at least one highly effective method of birth control for the duration of the study. This includes oral birth control pills, contraceptive implants, and intra-uterine devices. Diaphragms and condoms are not considered highly effective. Subjects not of reproductive potential will be exempt (e.g., post-menopausal, surgically sterilized)
9. If male, and partner is of childbearing potential, must be willing to utilize at least one highly effective method of birth control for the duration of the study. This includes oral birth control pills, contraceptive implants, and intra-uterine devices Diaphragms and condoms are not considered highly effective. Subjects not of reproductive potential will be exempt (surgically sterilized)

Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or intend to become pregnant during the study period.
2. Subjects whose caregivers are unable/unwilling to cooperate with the protocol requirements.
3. Subject will be excluded who are suffering with Rett syndrome and Childhood Disintegrative Disorder.
4. Other serious co-morbid medical disorders affecting brain function and behavior, including uncontrolled seizures.
5. Subjects unable to refrain from taking non-study antibiotics for the period of the study.
6. Subjects diagnosed with cancer, except small localized basal cell carcinoma.
7. Subjects known to abuse alcohol or drugs.
8. Subjects who have undergone gastric bypass or total colectomy, or who are scheduled for these procedures.
9. Infection with HIV.
10. Infection with Hepatitis B or C.
11. Allergy to benzodiazepine.
12. Inability to stop loperamide, diphenoxylatye/atropine, or cholestyramine before the study
13. Unable to stop opiate treatment unless on a stable dose including PRN dosing, and no dose increase planned for the duration of the study
14. Known positive stool cultures for enteropathogens including, but not limited to Shigella, Salmonella, and Campylobacter within 30 days before enrollment. (These infection agents should be treated in advance of participation in this FMT study because they affect the good flora).
15. Known stool studies positive for ova and/or parasites in 30 days prior to enrollment. (Same as above).
16. Planned travel outside United States during study period.
17. Hypersensitivity to vancomycin
18. Renal insufficiency
19. Colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
ATEC | 52 Weeks
  Number of participants with changes in the Autism Treatment Evaluation Checklist scores
QoLA | 52 Weeks
  Number of participants with changes in Quality of Life Autism scores
CARS-2 | 52 Weeks
  Number of participants with changes in Childhood Autism Rating Scale 2 scores
SRS-2 | 52 weeks
  Number of patients with changes in SRS-2 scores
Behavioral changes | 52 weeks
  Changes in reported incidence of disturbances in non-core aspects of behavior or function
GSRS | 52 weeks
  Number of patients with reported changes in GSRS measure of GI disturbances
abbrvCDAI | 52 weeks
  Number of patients with changes in abbrevCDAI scores
HSPP | 52 weeks
  Number of subjects with changes in quality of life metric HSPP

SECONDARY OUTCOMES:
Shannon Diversity Index | 52 Weeks
  Changes in Shannon Diversity index compared between pre and post FMT scores
Microbiome changes | 52 weeks
  Number of subjects with changes to microbiome relative abundance and composition

OTHER OUTCOMES:
Adverse Events | 52 Weeks
  Number of participants with grade III or higher adverse events
Serious Adverse Events | 52 Weeks
  Number of participants with serous adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Study Director — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No
HIPAA